CLINICAL TRIAL: NCT00690586
Title: Fluid Balance, Hormones and Urine Proteomics in Nephrotic Syndrome in Childhood
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: The Danish Medical Research Council (Other); The Danish Kidney Association (Other)
Responsible Party: Rene Frydensbjerg Andersen, Aarhus University Hospital
Other Study IDs: nsdk07-09
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2008-06

CONDITIONS: Nephrotic Syndrome
Keywords: Nephrotic syndrome; Underfill and overfill theory; Steroid resistance; Urine proteomics; AVP; ANP; Angiotensin II; Renin and Aldosterone
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples for hormone analyzes Urine samples for urine protomis, AQP II and ENaC
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to describe the hormones controlling fluid balance in pediatric patients with nephrotic syndrome. Further more, an analysis of the urinary and plasma proteins will be done using proteomics. Different composition of proteins in the urine or plasma might indicate if the patients will respond to treatment or not.

DETAILED DESCRIPTION:
Nephrotic syndrome represents the association of proteinuria, hypoalbuminemia, oedema and hyperlipidemia. The pathogenesis of the oedemas remains controversial. The "underfill" theory is the traditional explanation where massive proteinuria leads to low plasma albumine and a subsequent decrease in intravascular osmotic pressure leading to edema formations. Because most patients are normotensive and have normal intravascular pressure the "overfill" theory has been proposed suggesting a primary defect in renal sodium handling being responsible for oedema formation.

Ten percent of the children with nephrotic syndrome do not respond to standard steroid treatment and a significant proportion of these patients progress towards end-stage renal failure. At initial presentation it cannot be said if a patient will respond to treatment or not.

The purposes of the sudy:

1. To describe changes in the hormones, Aldosterone, Atrial Natriuretic Peptide (ANP), Arginin Vasopressin (AVP), Renin and Angiotensin II in patients with idiopathic nephrotic syndrome and to analyse to what extend the change in these hormones reflected a "underfill" or "overfill" situation.
2. To describe changes in the urine concentration of the water channel AQP II and the sodium channel ENaC during the course of nephrotic syndrome.
3. To test the hypothesis that urine and plasma proteomics from patients with steroid resistant nephrotic syndrome differs from patients with steroid sensitive nephrotic syndrome.

50 pediatric patients with nephrotic syndrome will be included after informed consent from both parents.

At day 1, 2, 3, 30 and 120 blood samples for hormones will be taken together with creatinin, albumine, Na+, K+, Hgb. An Echocardiography will be performed at day 1 and day 30 to determine v. cava inferior index.

At day 1,30 and 120 urine and plasma will be collected for proteomics and measurement of AQP II and ENaC concentrations.

Further more a clinical examination will be performed at day 1, 2, 3, 30 and 120 and weight, blood pressure and response to treatment will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Nephrotic syndrome, age below 15 years

Exclusion Criteria:

* Systemic disease e.g. Henoch-Schonleins purpura, Lupus erythematosus, diabetes mellitus
* Age over 15 years
* Treatment with diuretics prior to baseline blood samples

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with nephrotic syndrome will be included from 5 pediatric centrs in Denmark.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2007-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Søren Rittig, MD, Study Director — Aarhus University Hospital Skejby
Locations (1):
- Department of Pediatrics, Aarhus University Hospital, Skejby, Aarhus, Aarhus N, Denmark